CLINICAL TRIAL: NCT00916305
Title: Pilot Study of an Intervention Among Young People to Prevent Noise-induced Hearing Loss and Tinnitus
Brief Title: TUNE! Teaching the UK About Noise Exposure: A Pilot Study
Acronym: gildeaf1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Cambridge (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Clare Gilbert, Professor of International Eye Health, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Gilbert deafness 1
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Noise-induced Hearing Loss and Tinnitus
Keywords: deafness noise tinnitus hearingloss
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Tinnitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Audio video (Experimental): Participants will listen to an audio video modified to mimic noise induced hearing loss after one night at a loud club
  Interventions: Other: Modified Audio video
- Unmodified Audio video (Active Comparator): Participants will listen to the same music as the other arm, but only the track with unaltered music.
  Interventions: Other: Unmodified audio video

INTERVENTIONS:
Other: Modified Audio video — An audio video modified to mimic noise induced hearing loss after one night at a loud club
  Arms: Modified Audio video
Other: Unmodified audio video — An audio video with unaltered music
  Arms: Unmodified Audio video

SUMMARY:
In 1986 The Medical Research Council estimated that 4 million UK adolescents were at risk of hearing damage from over-exposure to loud music from personal audio players (PAPs), gigs, clubs, pubs and festivals. Since that time social noise exposure is estimated to have tripled to 19% of young people. The European Commission commissioned a report that estimated 5-10% of personal audio player users are risking permanent hearing loss and tinnitus by listening to music at high volumes for more than 1 hour a day for 5 years or more. Up to 246 million PAPs were sold in Europe in 2008, and 200 million mobile phones, many of which now have built-in audio players. Nevertheless, a recent survey showed that only 8% of young people identify hearing loss as a health problem. The Royal National Institute for the Deaf (RNID) undertook two surveys of young people in the UK to analyse listening behaviours as part of their "Don't Lose the Music" campaign. As a consequence they offer listening advice given by flyers at events and online at the dedicated website. There have been no studies to confirm if such advice is effective in reducing noise exposure.

Aim: This study will pilot a methodology for a randomised controlled trial to test the effectiveness of a publically-available online video in changing the listening habits of young music lovers i.e. reduce the volume and number of hours of exposure.

Hypothesis: A video and adapted sound track demonstrating the experience of noise-induced hearing loss and tinnitus accessed online will change the listening habits of 18-25 year-olds.

DETAILED DESCRIPTION:
Participants aged 18-25 years will be recruited by approaching staff at the LSHTM for recommendations of offspring or friends. Staff will be given information about the study and asked to provide an email address if the recruits are willing.

After obtaining informed consent online, participants will be randomized to active intervention i.e. an audio video demonstrating

* Normal hearing
* Temporary hearing damage after one night at a loud club
* Noise-induced hearing loss after repeated exposure (e.g. repeated clubbing for several months)
* Tinnitus related to noise exposure

Controls will watch the same video with an unaltered soundtrack.

Baseline data on listening habits and volumes will be collected prior to the intervention and again at 2 and 4 weeks. All data will be collected using an online system (survey monkey). At no point will researchers meet participants who will also not be known to each other.

Compliance will be assessed as participants will have to give a comment at the end of listening to the intervention.

Primary outcome: reduction is the proportion of time young people spend listening to music at a dangerous level i.e. equivalent to >80dB for 8 hours per day for 5 days a week

ELIGIBILITY:
Inclusion criteria:

* between 18 and 25 years of age
* used a portable listening device this year
* normal hearing
* no family history of hearing loss starting before 60 years of age

Exclusion criteria:

* recurrent or recent hearing loss, tinnitus or ear disease
* hearing loss beginning before 60 years of age in an immediate member of family

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Smith, MB ChB, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene and Tropical Medicine, London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 264 assessed for eligibility: 9 excluded 190 did not take initial survey - no reasons given
Period: Overall Study
Arm/Group | Modified Audio Video | Unmodified Audio Video
Started | 28 | 37
Completed | 7 | 9
Not Completed | 21 | 28
Not completed — Lost to Follow-up | 21 | 27
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Audio Video | Unmodified Audio Video | Total
Number analyzed (Participants) | 28 | 37 | 65
Age, Customized [Number; unit: participants]
  18-25 years | 28 | 37 | 65
Sex/Gender, Customized [Number; unit: Participants] — Per-arm data are not available. A total of 51 (78.5%) participants were female and a total of 14 (21.5%) participants were Male
  Participants
    Male/Female | 28 | 37 | 65

OUTCOME MEASURES:

1. Secondary Outcome: Reduction in Dangerous Listening Behaviour Defined as Daily Personal Noise Exposure in dB (LEPD) :to be Safe This Should Total Less Than 80dB
Description: Daily average over the previous month
Time Frame: 1 months
Measure: Mean (Standard Deviation); unit: Decibels per day
Arm/Group | Modified Audio Video | Unmodified Audio Video
Number analyzed (Participants) | 7 | 9
Decibels per day
  Baseline | 28 (31) | 58 (26)
  At 1 month | 32 (33) | 46 (15)

2. Primary Outcome: Reduction in Dangerous Listening Behaviour Defined as Weekly Personal Noise Exposure in dB (LEPD)
Description: Weekly average over the previous month
Time Frame: 1 months
Measure: Mean (Standard Deviation); unit: Decibels per week
Arm/Group | Modified Audio Video | Unmodified Audio Video
Number analyzed (Participants) | 7 | 9
Decibels per week
  Baseline | 71 (36) | 87 (16)
  At 1 month | 84 (40) | 79 (14)

ADVERSE EVENTS:
Description: Adverse events were not monitored in this study
Arm/Group | Modified Audio Video | Unmodified Audio Video
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No